CLINICAL TRIAL: NCT01882907
Title: An Open-label, Randomized, Active-controlled Study to Compare the Effect of 16 Weeks Treatment With Vildagliptin to Pioglitazone as add-on Therapy to Metformin in Type 2 Diabetic Patients Inadequately Controlled With Metformin Monotherapy
Brief Title: Safety and Efficacy Study to Compare Vildagliptin to Pioglitazone as Adding on Metformin in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237AKR05T
Record Dates: First submitted 2013-06-03; First posted 2013-06-21 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: Type 2 Diabetes
Keywords: vildagliptin; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vildagliptin (Experimental): vildagliptin add-on the therapy to metformin in patients with type 2 diabetes inadequately controlled with metformin monotherapy
  Interventions: Drug: vildagliptin
- pioglitazone (Active Comparator): Pioglitazone add-on the therapy to metformin in patients with type 2 diabetes inadequately controlled with metformin monotherapy
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: vildagliptin — vildagliptin 50mg bid for 16 weeks
  Other Names: Galvus
  Arms: vildagliptin
Drug: Pioglitazone — Pioglitazone 15mg bid for 16 weeks
  Other Names: Actos
  Arms: pioglitazone

SUMMARY:
The purpose of this study is to compare the effect of 16 weeks treatment with vildagliptin to pioglitazone as add-on the therapy to metformin in patients with type 2 diabetes inadequately controlled with metformin monotherapy.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a chronic progressive disease characterized by hyperglycemia that result from pancreatic islet dysfunction. Presently available oral antihypoglycemic drug improves glycemic control over the short term, none has been shown to stop the progressive decline in beta cell function which contributes to the deterioration of glycemic control over time.

Pathophysiology of T2DM is known as tissue resistance for insulin and progressive beta cell failure. Which one attributes first is unclear, but non-obese T2DM patients often show normal fasting plasma glucose (FPG) but postprandial plasma glucose (PPG) level is high and reduced or lacking normal compensatory insulin secretion. In Korea, more than 80% of T2DM are non-obese type (BMI >= 27 ) and it was observed that basal insulin level and compensatory insulin secretion reaction were reduced in normal healthy population. Based on that, metformin is an established first line treatment for type 2 diabetes, acting primarily to enhance hepatic and peripheral insulin sensitivity. However, it has become increasingly apparent that many patients require a combination of agents to attain optimal glycemic control.

Better understanding of incretin effect on the pathophysiology of T2DM has recently led to development of new oral hypoglycemic agents. Vildagliptin is a potent and highly selective dipeptidyl peptidase (DPP)-IV inhibitor that improves islet function by increasing pancreatic alpha and beta cell responsiveness to glucose. Studies in patients with T2DM have shown that vildagliptin significantly reduced HbA1c and FPG level from baseline and did not induce weight gain and the incidence of hypoglycemia was low. In addition, studies in rodents support an effort of vildagliptin on beta cell remodeling.

The thiazolidinediones are effective in reducing HbA1C in obese T2DM patients and it is known that only thiazolidinedione can delay the beta cell failure . But recently, thiazolidinediones were found to be associated with a decrease in bone mineral density and to raise the risk of myocardial infarct and cardiovascular related mortality. Thus, there is a need for new classes of blood glucose lowering drug which has the potential to delay or prevent the progression of T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Age in the range of 18 to 80 years
2. HbA1c 7 to 11%
3. FPG < 270 mg/dL (15 mmol/L);
4. Agreement to maintain prior diet & exercise
5. Written informed consent to participate in the study

Exclusion criteria:

1. Type 1 diabetes or Any kind of secondary diabetes
2. Pregnant or lactating women
3. Acute infections which may affect blood glucose control within 4 weeks prior to visit 1.
4. Significant diabetes complications e.g., symptomatic autonomic neuropathy or gastroparesis
5. Previous history of severe cardiovascular disease such as

   1. Torsades de Pointes, sustained and clinically relevant ventricular tachycardia, or ventricular fibrillation
   2. Percutaneous coronary intervention within the past 3 months
6. Any of the following within the past 6 months

   1. Myocardial infarction (MI) (if the visit 1 ECG reveals patterns consistent with an MI and the date of the event cannot be determined, then the patient can enter the study at the discretion of the investigator and the sponsor)
   2. Coronary artery bypass surgery
   3. Unstable angina
   4. Stroke
7. Congestive heart failure (NYHA class I to IV)
8. Liver disease such as cirrhosis or chronic active hepatitis
9. Known sensitivity to pioglitazone, rosiglitazone, or similar drugs
10. Chronic insulin treatment (> 4 weeks of treatment in the absence of an intercurrent illness) within the past 6 months
11. Chronic oral or parenteral corticosteroid treatment (> 7 consecutive days of treatment) within 8 weeks prior to visit 1
12. Any of the following laboratory abnormalities

    1. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) greater than 2.5 times the upper limit of the normal range at visit 1
    2. Direct bilirubin greater than 1.3 times the upper limit of the normal range at visit 1
    3. Serum creatinine levels > 2.5 mg/dL (220 μmol/L) at visit 1
    4. Clinically significant thyroid-stimulating hormone (TSH) outside normal range at visit 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In Ju Kim, MD, Principal Investigator — Pusan National University Hospital
Locations (15):
- South Korea (15):
  - Busan Saint Mary's Medical Center, Busan
  - Dong-AUniversity Medical Center, Busan
  - Inje University Baik Hospital, Busan
  - Kosin University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Changwon Fatima Hospital, Changwon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungbuk National Universtiy Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Masan Samsung Medical Center, Masan
  - Ulsan University Hospital, Ulsan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total number of patients who were in screening is 287. However, 59 patients were excluded. 49 Patients didn't meet inclusion/exclusion criteria. 10 Patients didn't take investigational product.
  As a result, 228 patients took investigational product.
Period: Overall Study
Arm/Group | Vildagliptin | Pioglitazone
Started (The patients who were screening failure and didn't taking investigational product are excluded.) | 117 | 111
Completed | 103 | 83
Not Completed | 14 | 28
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 0 | 3
Not completed — Lost to Follow-up | 1 | 4
Not completed — Protocol Violation | 10 | 14
Not completed — Withdrawal by Subject | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vildagliptin | Pioglitazone | Total
Number analyzed (Participants) | 117 | 111 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.8) | 53.9 (9.1) | 54.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 63 | 130
  Male | 50 | 48 | 98
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 24.9 (3.2) | 25.0 (3.3) | 24.9 (3.3)
Duration of diaebetes [Mean (Standard Deviation); unit: months] | 68.3 (62.0) | 60.2 (58.6) | 64.3 (60.4)

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of HbA1C Change From Baseline in Vildagliptin + Metformin Group Compared With Pioglitazone + Metformin Group
Time Frame: 16 weeks
Population: This number is analyzed subjects population(Vildagliptin group n=115, Pioglitazone group n=108). It is excluded the patients who are screening failure and not available to efficacy assessment.
Measure: Mean (Standard Deviation); unit: % (change of HbA1c)
Arm/Group | Vildagliptin | Pioglitazone
Number analyzed (Participants) | 115 | 108
% (change of HbA1c) | -0.94 (0.79) | -0.60 (1.12)

2. Secondary Outcome: the Mean Changes of FPG and PPG From Baseline Between Vildagliptin + Metformin and Pioglitazone + Metformin Groups
Description: 1. After 16 weeks, to assess the effect of vildagliptin compared with the effect of pioglitazone on Fasting Plasma Glucose (FPG)
  2. After 16 weeks, to assess the effect of vildagliptin compared with the effect of pioglitazone on Postprandial Glucose (PPG)
Time Frame: 16 weeks , visit 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Vildagliptin: vildagliptin add-on the therapy to metformin in patients with type 2 diabetes inadequately controlled with metformin monotherapy
  vildagliptin: vildagliptin 50mg bid for 16 weeks
  The mean changes in FPG from baseline to week 16 were -20.4 mg/dL The mean changes in PPG levels from baseline to week 16 were -60.2 mg/dL
- Pioglitazone: Pioglitazone add-on the therapy to metformin in patients with type 2 diabetes inadequately controlled with metformin monotherapy
  Pioglitazone: Pioglitazone 15mg bid for 16 weeks
  The mean changes in FPG from baseline to week 16 were -15.0 mg/dL The mean changes in PPG levels from baseline to week 16 were -38.2 mg/dL
Arm/Group | Vildagliptin | Pioglitazone
Number analyzed (Participants) | 115 | 108
mg/dL
  FBG levels difference | -20.41 (34.81) | -15.04 (38.15)
  PPG levels difference | -60.23 (75.48) | -38.19 (83.79)

3. Secondary Outcome: the Mean Changes of Lipid Profiles From Baseline Between Vildagliptin + Metformin and Pioglitazone + Metformin Groups
Description: The Mean Changes of Lipid Profiles(Triglyceride, Total cholesterol, LDL, HDL, Non-HDL cholesterol) From Baseline Between Vildagliptin + Metformin and Pioglitazone + Metformin Groups after 16weeks
Time Frame: 16 weeks, visit 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vildagliptin | Pioglitazone
Number analyzed (Participants) | 115 | 108
mg/dL
  Triglyceride | -9.22 (55.98) | -4.79 (67.83)
  Total cholesterol | -6.45 (25.10) | 9.60 (33.83)
  LDL | -6.03 (21.20) | 5.38 (30.37)
  HDL | -0.34 (8.57) | 3.69 (10.33)
  Non-HDL cholesterol | -8.39 (24.67) | 5.79 (32.72)

4. Secondary Outcome: the Mean Changes of Body Weight From Baseline Between Vildagliptin + Metformin and Pioglitazone + Metformin Groups
Time Frame: 16 weeks, visit 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Vildagliptin | Pioglitazone
Number analyzed (Participants) | 115 | 108
kg | -0.07 (1.53) | 0.69 (2.07)

5. Secondary Outcome: the Mean Changes of Insulin, C-peptide, HOMA-IR, HOMA-beta From Baseline Between Vildagliptin + Metformin and Pioglitazone + Metformin Groups
Time Frame: 16 weeks, visit 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcU/mL*mmol/L
Arm/Group | Vildagliptin | Pioglitazone
Number analyzed (Participants) | 115 | 108
mcU/mL*mmol/L
  Insulin difference | 0.36 (6.95) | -8.21 (70.06)
  C-peptide difference | 0.07 (0.84) | -0.24 (1.14)
  HOMA-IR difference | -0.06 (2.92) | -3.33 (25.16)
  HOMA-beta difference | 9.77 (28.10) | -24.26 (294.88)

6. Other Pre Specified Outcome: the Numbers of Participants With Adverse Events Between Vildagliptin + Metformin and Pioglitazone + Metformin Groups
Time Frame: 16 weeks, visit 3,4,5
Population: This number is subject population who were exposure the drug(Vildagliptin group n=117, Pioglitazone group n=111). It is excluded the patients who are screening failure.
Measure: Number; unit: participants
Arm/Group | Vildagliptin | Pioglitazone
Number analyzed (Participants) | 117 | 111
participants
  Number of incidence | 27 | 25
  Number of adverse events | 48 | 37

ADVERSE EVENTS:
Arm/Group | Vildagliptin | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 4/117 | 2/111
Other Adverse Events (participants affected / at risk) | 16/117 | 11/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vildagliptin (N=117) | Pioglitazone (N=111)
Urinary tract infection (Immune system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Injury of ligament (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Upper respiration infection (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vildagliptin (N=117) | Pioglitazone (N=111)
Common cold (Infections and infestations) | 3 | 4
Upper respiration infection (Infections and infestations) | 4 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dizziness (Nervous system disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days